CLINICAL TRIAL: NCT05894291
Title: Evaluation Two Different Prone Position Techniques on the Occurrence of Pressure Sores in Patients With Invasive Mechanical Ventilation With Acute Respiratory Distress Syndrome in the Intensive Care Unit : a Multicenter, Prospective Randomized Controlled Trial.
Brief Title: Comparaison of Two Prone Position Techniques on Occurence of Pressure Sores in ICU
Acronym: PROPOSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: UNIVERSITY HOSPITAL, ORLEANS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DR220257/PROPOSE; IDRCB (Registry Identifier: 2022-A02601-42)
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Acute Respiratory Distress Syndrome; Pressure Ulcers Stage III
Keywords: ARDS; Pressure Sores; Pressure Ulcer; Acute Respiratory Distress Syndrome; Prone Position; Swimmer Position
MeSH Terms: conditions — Respiratory Distress Syndrome; Pressure Ulcer | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swimmer Prone Position (Experimental)
  Interventions: Other: Swimmer Prone Position
- Prone position with arms alongside the body (Active Comparator)
  Interventions: Other: Prone position with arms alongside the body

INTERVENTIONS:
Other: Swimmer Prone Position — Patients will be positioned with the head rotated. This rotation is followed by shoulder elevation/abduction, then 90° elbow flexion for the arm opposite to the head rotation. The hand is placed flat on the bed.
  A 60° to 90° flexion is performed on the hip homolateral to head rotation, combined with knee flexion.
  The position is changed to the mirror position every 4 hours.
  Arms: Swimmer Prone Position
Other: Prone position with arms alongside the body — The head will be positioned either straight or rotated to one side, depending on ICU habits. The arms are positioned symmetrically along the body, palms up. The lower limbs are positioned symmetrically and parallel, knees extended or slightly flexed if a cushion is used on the front of the feet.
  Head rotation, if applicable, is performed every 4 hours.
  Arms: Prone position with arms alongside the body

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a diffuse inflammation of the lungs that occurs in a variety of diseases. According to the Berlin definition, ARDS is characterized by diffuse lung damage in patients with predisposing factors. Understanding the physiology of ARDS has led to improved ventilatory management, which must be protective to ensure adequate oxygenation and CO2 clearance. Prone position (PP) is a technique that can reduce mortality in patients with severe ARDS. PP results in a more homogeneous distribution of pulmonary stress and strain, helping to protect the lung against ventilator-induced lung injury (VILI). It also increases the PaO2/FiO2 (P/F) ratio, improves the pulmonary ventilation-perfusion ratio, decreases PaCO2 and promotes ventilation of the dorsal lung regions. This technique should be offered to all patients with severe ARDS for 16 consecutive hours, to improve survival and weaning success from mechanical ventilation. However, PP has adverse effects. A meta-analysis showed an increased risk of pressure sores, possibly linked to generalized acute inflammation associated with significant cytokine discharge and diffuse lesions of the vascular endothelium. PP also increased the risk of obstruction and displacement of the endotracheal tube. Final positioning in PP, (i.e., the position imposed on the patient for the duration of the PP session) varies from one ICU to another, and is rarely described in scientific articles. There are two main variants:

1. prone , with arms alongside the body
2. prone, swimmer's position

The aim of our study is to show that the "swimmer" PP reduces the occurrence of stage 3 or higher pressure sores, compared with the "arms alongside the body" PP (standard care) at Day 28 post inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Intubated patient on invasive mechanical ventilation with moderate to severe acute respiratory distress syndrome according to the BERLIN classification with a P/F ratio < 150, requiring prone position.
* Express consent of the patient or representative or in the absence of this, emergency inclusion procedure
* Health insurance coverage

Exclusion Criteria:

* Patient with 2 (or more) Prone position sessions
* Patient in whom one of the two positions could not be achieved: (Joint limitation; Neck size that would prevent head rotation; Orthopaedic spinal or segmental trauma; BMI greater than 45)
* Presence of stage 2 or higher pressure ulcers on the anterior parts of the body at screening
* Presence of extracorporeal membrane oxygenation (ECMO)
* Patient already included in the study
* Pregnant or breastfeeding woman
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of stage 3 or higher pressure ulcers | Day 28 after randomization
  Percentage of patients who acquired at least one stage 3 or 4 pressure ulcer between day 1 (randomization) and day 28 according to the revised pressure injury staging system (Edsberg, J Wound Ostomy Cont Nurs, 2016). Death and resolution of ARDS will be considered as events in competition with the occurrence of a Stage 3 or higher pressure ulcer.

SECONDARY OUTCOMES:
Mortality at day 28 | Day 28 after randomization
  Mortality rate at day 28
In-hospital Mortality at day 90 | Day 90 after randomization
  In-hospital Mortality rate at day 90
Number of days without mechanical ventilation at D28 | Day 28 after randomization
  Ventilator Free days at day 28
Length of stay in intensive care unit (censored at Day 90) | Day 90 after randomization
  Length of stay in intensive care unit after randomization (censored at D90)
Length of hospital stay (censored at D90) | Day 90 after randomization
  Length of hospital stay after randomization (censored at D90)
Presence of ICU acquired weakness at discharge from ICU | Day 28 after randomization
  Rate of patients with ICU acquired weakness defined by MRC score less than 48 at ICU discharge
Occurrence of scapulohumeral joint dislocation during prone period | Day 28 after randomization
  Number of patients with at least one radiologically proven scapulohumeral dislocation during a prone position period

CONTACTS AND LOCATIONS:
Locations (1):
- UHT of Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Labeau SO, Afonso E, Benbenishty J, Blackwood B, Boulanger C, Brett SJ, Calvino-Gunther S, Chaboyer W, Coyer F, Deschepper M, Francois G, Honore PM, Jankovic R, Khanna AK, Llaurado-Serra M, Lin F, Rose L, Rubulotta F, Saager L, Williams G, Blot SI; DecubICUs Study Team; European Society of Intensive Care Medicine (ESICM) Trials Group Collaborators. Prevalence, associated factors and outcomes of pressure injuries in adult intensive care unit patients: the DecubICUs study. Intensive Care Med. 2021 Feb;47(2):160-169. doi: 10.1007/s00134-020-06234-9. Epub 2020 Oct 9. PMID 33034686
- [Background] Girard R, Baboi L, Ayzac L, Richard JC, Guerin C; Proseva trial group. The impact of patient positioning on pressure ulcers in patients with severe ARDS: results from a multicentre randomised controlled trial on prone positioning. Intensive Care Med. 2014 Mar;40(3):397-403. doi: 10.1007/s00134-013-3188-1. Epub 2013 Dec 19. PMID 24352484
- [Background] Sud S, Friedrich JO, Taccone P, Polli F, Adhikari NK, Latini R, Pesenti A, Guerin C, Mancebo J, Curley MA, Fernandez R, Chan MC, Beuret P, Voggenreiter G, Sud M, Tognoni G, Gattinoni L. Prone ventilation reduces mortality in patients with acute respiratory failure and severe hypoxemia: systematic review and meta-analysis. Intensive Care Med. 2010 Apr;36(4):585-99. doi: 10.1007/s00134-009-1748-1. Epub 2010 Feb 4. PMID 20130832